CLINICAL TRIAL: NCT05611359
Title: Resection of the Primary Pancreatic Tumour and Thermal Hepatic Ablation Combined With Chemotherapy vs. Chemotherapy in Hepatic Oligometastatic Pancreatic Cancer: A Randomized Controlled Trial
Brief Title: Surgery and Thermal Hepatic Ablation Combined With Chemotherapy in Hepatic Oligometastatic Pancreatic Cancer
Acronym: HOPE-1
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0698
Record Dates: First submitted 2022-11-06; First posted 2022-11-10 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Pancreatic Ductal Adenocarcinoma
Keywords: Pancreatic Ductal Adenocarcinoma; Hepatic Metastasis; Thermal Ablation
MeSH Terms: interventions — Transurethral Resection of Prostate; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thermal Ablation (Experimental): In the patients with liver oligometastasis after pancreatic ductal adenocarcinoma (PDAC) surgery, thermal ablation and chemotherapy are administered.
  Interventions: Procedure: Thermal Ablation; Drug: Chemotherapy
- Chemotherapy (Active Comparator): In the patients with liver oligometastasis after pancreatic ductal adenocarcinoma (PDAC) surgery, chemotherapy is administered.
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Procedure: Thermal Ablation — Thermal hepatic ablation Combined with Chemotherapy
  Other Names: Thermal Ablation Combined with Chemotherapy
  Arms: Thermal Ablation
Drug: Chemotherapy — Chemotherapy

SUMMARY:
The goal of this clinical trial is to compare the overall survival of thermal ablation combined with chemotherapy and chemotherapy alone in the patients with liver oligometastasis after pancreatic ductal adenocarcinoma (PDAC) surgery.

The main question it aims to answer is: whether thermal ablation combined with chemotherapy can effectively prolong the overall survival in the patients with liver oligometastasis after pancreatic ductal adenocarcinoma (PDAC) surgery.

The participants in the treatment group will receive systemic chemotherapy combined with liver thermal ablation, while the participants in the control group will receive chemotherapy alone. All participants will be followed up to evaluate the overall survival after treatment.

DETAILED DESCRIPTION:
How to improve the overall survival in the patients with liver oligometastasis after pancreatic ductal adenocarcinoma (PDAC) surgery is still a huge challenge in clinic. Chemotherapy is still the first-line treatment for patients with liver oligometastasis after PDAC resection. On the basis of chemotherapy, the clinical benefits of removing hepatic oligometastasis by thermal ablation are still unclear. In this study, we will recruit patients with liver oligometastasis after PDAC surgery to explore the effect of thermal ablation combined with chemotherapy on the overall survival of patients.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age ≥ 18; (2) pancreatic ductal adenocarcinoma was confirmed by pathology; (3) The patient's liver function was Child Pugh A or B ; (4) Karnofsky score ≥ 80; (5) There is a safe puncture path under the guidance of ultrasound for liver oligometastatic tumor; (6) Single diameter of liver oligometastatic tumor ≤ 5 cm, or ≤ 3 liver oligometastatic tumors, each diameter ≤ 3 cm; (7) Platelet count>40000/mm3; (8) Thrombin time ratio>40%; (9) Sign the Informed Consent of Clinical Trial.

Exclusion Criteria:

* (1) Refuse to receive chemotherapy or thermal ablation; (2) >3 liver metastases or extrahepatic metastases (such as peritoneum, lung, bone or brain); (3) Single diameter of liver oligometastatic tumor>5 cm; (4) The patient has ascites, portal vein thrombosis, or bile duct dilatation or stenosis; (5) Presence of another malignant tumors; (6) Prior anti-tumor treatment (including radiotherapy, chemotherapy and thermal ablation); (7) Presence of central nervous system abnormalities, mental diseases, unstable angina, congestive heart failure, serious arrhythmia or other serious diseases; (8) Use of anticoagulants maintenance treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 2 years
  Time from enrollment to death

SECONDARY OUTCOMES:
Progression-free survival time | 2 years
  Time from thermal ablation to recurrence of liver lesion
Procedure related complications | up to 12 months
  Relevant complication after thermal ablation
Procedure related mortality | up to 12 months
Patient satisfaction | 2 years
  Satisfaction questionnaire designed by investigator group
Medical cost | 2 years
  Hospital expenditure
Serum concentration of serological examinationof liver function | 2 years
  Serum concentration of tunmor biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: pintong huang, Doctor, Study Chair — the 2th affiliated hospital of zhejiang university school of medicine

IPD SHARING:
Plan to Share IPD: No